CLINICAL TRIAL: NCT07078851
Title: Comparing the Efficacy and Safety of Fractional Picosecond Laser and Gold Microneedle in the Treatment of Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jin Chen, Chief Physician, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 500103014
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acne Scarring; Acne Scars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Picosecond Laser Group (Experimental)
  Interventions: Device: Fractional Picosecond Laser Treatment
- gold microneedle group (Experimental)
  Interventions: Device: gold microneedle treatment

INTERVENTIONS:
Device: Fractional Picosecond Laser Treatment — Compound lidocaine cream (Tongfang Pharmaceutical Group Co., Ltd., National Drug Approval Number: H20063466) was applied to the face. After 60 minutes, it was cleaned thoroughly in preparation for treatment. The subjects lay flat on the treatment bed, and the face was disinfected twice. Treatment was performed using the Picsure Focus Lens (Cynosure, USA, Registration Certificate Number: National Medical Device Import 20153242702) with the following parameters: 6mm spot size, focus filter, 755nm wavelength, energy of 6.0J/cm², and 2Hz frequency. The endpoint response was skin flushing and mild edema. Immediately after the operation, recombinant human epidermal growth factor (Kanghesu, 20000IU/4ml/vial, Shanghai Haohai Biological Technology Co., Ltd.) was applied externally, followed by wet compresses with saline gauze combined with cold spray for 30 minutes. The subjects were required to apply recombinant human epidermal growth factor to the entire facial skin twice a day (one vial each
  Arms: Fractional Picosecond Laser Group
Device: gold microneedle treatment — The face was topically anesthetized with compound lidocaine cream (Tongfang Pharmaceutical Group Co., Ltd., National Drug Approval No. H20063466). After 60 minutes, the cream was cleaned off thoroughly to prepare for treatment. The subject was positioned supine on the treatment bed, and the face was disinfected twice. Gold microneedle radiofrequency treatment was performed using the NDPRD00009-E 3DEEP Phased RF治疗仪 (Eedy Med, Israel). The gold microneedle handpiece was disinfected with 95% medical ethanol. Under sterile conditions, the microneedle tips were installed, and the treatment parameters were set as follows: Cheeks mode with Intensif method, microneedle length 0.8-2.0 mm (length <1.5 mm for forehead, temporal region, and zygomatic bone prominences); RF output time 180 ms; RF power 6-16 W. The operator held the device vertically and applied it evenly across the treatment area in a grid pattern, ensuring gentle contact with the skin to avoid excessive pressure. Any untreated gaps
  Arms: gold microneedle group

SUMMARY:
The goal of this clinical trial is to compare a 755nm honeycomb picosecond laser versus a CO2 fractional laser for the treatment of atrophic acne Efficacy and safety of scarring.

The main questions it aims to answer are:

Effectiveness of 755nm Honeycomb Picosecond Laser and CO2 Fractional Laser in the Treatment of Atrophic Acne Scars

Effectiveness of scarring

Participants will:

the control group(receiving 10600nm CO₂ fractional laser[AFL]treatment)and the experimental group(receiving picosecond laser with honeycomb focusing lens array[P-DLA]treatment).Facial images were captured using the VISIA skin imaging system,and the red zone,UV spot,and brown spot scores were evaluated for all subjects before each treatment,and at 1 and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with symmetrical atrophic acne scars on both sides of the face by a dermatologist; 2）Age ≥ 18 years old; 3) Voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. History of scar tissue in the past The person; 2) History of phototherapy such as laser and radiofrequency in the past 3 months; 3) History of photosensitivity or within the past 3 months Individuals who have taken photosensitive drugs; 4) Individuals allergic to lidocaine; 5) Individuals with coagulation dysfunction; 6) In the past 3 months History of oral corticosteroids and immunosuppressants; 7) Malignant tumor patients; 8) During pregnancy or lactation Women; 9) Individuals with local facial infections or injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
ECCA score | 0, 4, 8, 12, 16, 24 weeks
  Echelle d 'Evaluation Clinique des Cicatrices d 'acne

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided